CLINICAL TRIAL: NCT06793254
Title: Translation, Cultural Adaptation and Validation of the Italian Version of Functional Rating Index in Patients With Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Salvatore Simone Vullo, MD, Doctor, Azienda Ospedaliera Brotzu
Other Study IDs: I-FRI
Record Dates: First submitted 2025-01-19; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: This is a non-interventional study — None (this is a non-interventional study)

SUMMARY:
Chronic Low Back Pain (cLBP) is a global health issue lasting more than 3 months, where a clear pathologic and anatomic cause of pain is not recognized. Various personal and psychosocial factors can influence the onset and chronicity of low back pain.

The Functional Rating Index (FRI) is a self-administered questionnaire composed by 10 items, scored from 0 (better condition) to 4 (worst condition), that evaluate pain, sleep, work and daily activity. The FRI's final score ranges from 0% to 100% (no disability to severe disability). The aim of the study is to translate, culturally adapt and validate the FRI in Italian (I-FRI).

DETAILED DESCRIPTION:
Chronic Low Back Pain (cLBP) is a global health issue lasting more than 3 months, where a clear pathologic and anatomic cause of pain is not recognized. Various personal and psychosocial factors can influence the onset and chronicity of low back pain. An outcome measure, in a specific context, refers to a quantifiable or observable variable used to assess and evaluate the results or effects of a particular intervention, treatment, program, or research study. The choice of appropriate outcome measures is critical in research and evaluation because it directly influences the validity and reliability of the results. There are already other validated scales translated in Italian for the evaluation of patients with cLBP, such as the Oswestry Disability Index (ODI-I). The Functional Rating Index (FRI) is a self-administered questionnaire composed by 10 items, scored from 0 (better condition) to 4 (worst condition), that evaluate pain, sleep, work and daily activity. The FRI's final score ranges from 0% to 100% (no disability to severe disability).

The aim of the study is to translate, culturally adapt and validate the FRI in Italian (I-FRI). 104 patients were recruited for this study following inclusion/exclusion criteria. After signing the informed consent, each participant completed I-FRI, Oswestry Disability Index (ODI), Tampa Scale of Kinesiophobia (TSK) and Pain Catastrophizing Scale (PCS). All the patients have done the I-FRI re-test after 7 days from the first test administration.

All statistical analyses have been performed using IBM-SPSS (Statistical Package for the Social Sciences) version 23.00.

The results have been analyzed through the calculation of the Cronbach's alpha, the Intraclass Correlation Coefficient (ICC) and the Pearson's correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low Back Pain
* Adult age
* Reading/speaking Italian.

Exclusion Criteria:

* Acute low back pain (lasting up to 4 weeks) or subacute low back pain (lasting up to 12 weeks).
* Cognitive impairment.
* Disabling pathological conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with chronic low back pain
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-01-19 (Actual)

PRIMARY OUTCOMES:
Italian Version of Functional Rating Index (I-FRI) | Baseline
  self-administered questionnaire composed by 10 items, scored from 0 (better condition) to 4 (worst condition), that evaluate pain, sleep, work and daily activity. The FRI's final score ranges from 0% to 100% (no disability to severe disability).
Italian Version of Functional Rating Index (I-FRI) | After 7-10 days later the first assessment (please, see above) as concerns test-retest assessment reliability.
  self-administered questionnaire composed by 10 items, scored from 0 (better condition) to 4 (worst condition), that evaluate pain, sleep, work and daily activity. The FRI's final score ranges from 0% to 100% (no disability to severe disability).

SECONDARY OUTCOMES:
ODI (Oswestry Disability Index) | Baseline
  Oswestry Disability Index; score varying from 0 to 50, with higher scores indicating greater disability
PCS (Pain Catastrophizing Scale) | Baseline
  Pain Catastrophizing Scale; score varying from 0 to 52, with higher scores indicating greater catastrophizing
pain NRS (Numerical pain Rating Scale) | Baseline
  Numerical pain Rating Scale; score varying from 0 to 10, with higher scores indicating greater pain intensity
TSK (Tampa Scale of Kinesiophobia) | Baseline
  This self-report questionnaire assesses fear-avoidance behaviors. The investigators used the Italian 13-item version, with the reversed items removed, which has proven to be reliable and valid. Each item is scored using a four-point Likert scale, ranging from 1 (strongly disagree) to 4 (strongly agree). The total score is calculated by summing the individual item scores (range 13-52), with higher scores indicating greater kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Simone Vullo, Principal Investigator — Dottor
Locations (1):
- Salvatore Simone Vullo, Cagliari, Sardinia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clark S, Horton R. Low back pain: a major global challenge. Lancet. 2018 Jun 9;391(10137):2302. doi: 10.1016/S0140-6736(18)30725-6. Epub 2018 Mar 21. No abstract available. PMID 29573869
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Dagenais S, Caro J, Haldeman S. A systematic review of low back pain cost of illness studies in the United States and internationally. Spine J. 2008 Jan-Feb;8(1):8-20. doi: 10.1016/j.spinee.2007.10.005. PMID 18164449
- [Background] Makris UE, Higashi RT, Marks EG, Fraenkel L, Gill TM, Friedly JL, Reid MC. Physical, Emotional, and Social Impacts of Restricting Back Pain in Older Adults: A Qualitative Study. Pain Med. 2017 Jul 1;18(7):1225-1235. doi: 10.1093/pm/pnw196. PMID 27516362
- [Background] Feise RJ, Michael Menke J. Functional rating index: a new valid and reliable instrument to measure the magnitude of clinical change in spinal conditions. Spine (Phila Pa 1976). 2001 Jan 1;26(1):78-86; discussion 87. doi: 10.1097/00007632-200101010-00015. PMID 11148650
- [Background] Monticone M, Giorgi I, Baiardi P, Barbieri M, Rocca B, Bonezzi C. Development of the Italian version of the Tampa Scale of Kinesiophobia (TSK-I): cross-cultural adaptation, factor analysis, reliability, and validity. Spine (Phila Pa 1976). 2010 May 20;35(12):1241-6. doi: 10.1097/BRS.0b013e3181bfcbf6. PMID 20216338
- [Background] Monticone M, Baiardi P, Ferrari S, Foti C, Mugnai R, Pillastrini P, Rocca B, Vanti C. Development of the Italian version of the Pain Catastrophising Scale (PCS-I): cross-cultural adaptation, factor analysis, reliability, validity and sensitivity to change. Qual Life Res. 2012 Aug;21(6):1045-50. doi: 10.1007/s11136-011-0007-4. Epub 2011 Sep 13. PMID 21912846
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561